CLINICAL TRIAL: NCT02568553
Title: A Phase I Trial of the Combination of Lenalidomide and Blinatumomab in Patients With Relapsed or Refractory Non-Hodgkins Lymphoma (NHL)
Brief Title: Lenalidomide and Blinatumomab for the Treatment of Relapsed Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01640; NCI-2015-01640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-79; 9924 (Other: City of Hope Comprehensive Cancer Center LAO); 9924 (Other: CTEP); UM1CA186644 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Burkitt Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Recurrent Grade 3b Follicular Lymphoma; Recurrent Gray-Zone Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mediastinal Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Burkitt Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Grade 1 Follicular Lymphoma; Refractory Grade 2 Follicular Lymphoma; Refractory Grade 3 Follicular Lymphoma; Refractory Grade 3a Follicular Lymphoma; Refractory Gray-Zone Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Mediastinal Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (blinatumomab, lenalidomide) (Experimental): INDUCTION: Patients receive blinatumomab IV continuously on days 1-56 and lenalidomide PO on days 29-49 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients achieving response including stable disease receive blinatumomab IV continuously on days 1-7 and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receiving response including stable disease after completion of Consolidation receive lenalidomide PO on days 1-21. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Blinatumomab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide and blinatumomab when given together in treating patients with non-Hodgkin lymphoma that has returned after a period of improvement (relapsed). Biological therapies, such as lenalidomide, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Blinatumomab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of lenalidomide when given in combination with blinatumomab in the proposed regimen.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity anti-tumor response (complete response [CR] and partial response [PR] as per International workshop lymphoma response criteria).

II. To investigate the immune response to blinatumomab alone and in combination with lenalidomide.

III. To document the infection rate with a 96-hour bag change schedule for blinatumomab.

OUTLINE: This is a dose-escalation study of lenalidomide.

INDUCTION: Patients receive blinatumomab intravenously (IV) continuously on days 1-56 and lenalidomide orally (PO) on days 29-49 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients achieving response including stable disease receive blinatumomab IV continuously on days 1-7 and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receiving response including stable disease after completion of Consolidation receive lenalidomide PO on days 1-21. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed relapsed cluster of differentiation (CD)19+ non-Hodgkin lymphoma (NHL) (included in this category are follicular grade I, II, III, marginal zone, mantle cell, gray zone, primary mediastinal, Burkitt's, diffuse large B cell, small lymphocytic lymphoma); patients previously treated with CD19-targeted therapy (including chimeric antigen receptor T-cells [CAR T]) must have a subsequent biopsy and/or flow cytometry confirming CD19 positivity
* Karnofsky >= 60%
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count > 1000/mcL
* Platelets >= 50,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* AST (SGOT)/ALT(SGPT) (only if elevated liver function tests [LFTs] are due to disease) =< 5.0 x institutional upper limit of normal
* Body surface area (BSA)-normalized creatinine clearance >= 60 mL/min/1.73 m^2 (using Cockcroft-Gault creatinine clearance [CrCl])
* Patients must have had at least two prior chemotherapeutic or biologic (e.g. rituximab alone) regimens and not currently eligible for standard curative options; steroids alone and local radiation do not count as regimens; radiation to > 1 site and transplant are considered prior regimens
* Any prior therapy must have been completed at least 4 weeks prior to entry into the study
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Patients must have radiographically measurable disease; radiographically measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan; lesions in previously irradiated anatomic areas (external beam radiation) cannot be considered target lesions unless there has been documented growth of those lesions after radiotherapy
* Ability to understand and the willingness to sign a written informed consent document
* Human immunodeficiency virus (HIV) infected patients are eligible provided they meet all the other eligibility criteria of the study in addition to the following:

  * During prior lymphoma therapy, patients must not have experienced documented infections attributed to the HIV+ status
  * No history of non-adherence to cART and willing to adhere to cART while on study
  * Antiretroviral drugs with overlapping or similar toxicity profiles as study agents not allowed:

    * Efavirenz not allowed due to potential central nervous system (CNS) toxicity
    * Stavudine not allowed due to potential neuropathic effects
    * Zidovudine not allowed due to myelosuppressive effects
  * Patients must be willing to be followed at a minimum of approximately every 3 months by physician expert in HIV disease management
* Patients must be willing to be followed at a minimum of approximately every 3 months by physician expert in HIV disease management

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide and blinatumomab or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because lenalidomide is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known active hepatitis, type B or C; patients on suppressive therapy with a negative viral load and no evidence of hepatic damage are eligible
* Prior treatment with lenalidomide within 8 weeks prior to entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity | Up to 24 months
  Will be graded as according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 beginning April 1, 2018). Toxicities (grade, type, cycle, and attribution) experienced will be listed for each patient and summarized using standard descriptive methods.

SECONDARY OUTCOMES:
Clinical anti-tumor response (complete response and partial response as per International workshop lymphoma response criteria) | Up to 24 months
  Will be summarized using standard descriptive methods.
Changes in the frequency of CD4+ T cells | Baseline to up to day 57
  Will be assessed and compared at each time point, using regression methods that incorporate repeated measures. For each of the first 2 CD4+ measures, will compare the day 0 values (prior to any treatment) to the day 15 values (after 2 weeks of blinatumomab) and the day 57 (after 4 weeks of the both blinatumomab and lenalidomide) to the day 15 value. Additional analysis, will be undertaken to explore the relationship between changes (or lack of changes) and response. The paired-sample t-test will be used to provide a sense of the power/sensitivity that will be available for these comparisons.
Changes in the production of interferon (INF)-gamma from CD4+ T cells | Baseline to up to day 57
  Will be assessed and compared at each time point, using regression methods that incorporate repeated measures. For each of the first CD8+ T-cell frequencies and INF-gamma production, will compare the day 0 values (prior to any treatment) to the day 15 values (after 2 weeks of blinatumomab) and the day 57 (after 4 weeks of the both blinatumomab and lenalidomide) to the day 15 value. Additional analysis, will be undertaken to explore the relationship between changes (or lack of changes) and response. The paired-sample t-test will be used to provide a sense of the power/sensitivity that will be available for these comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (24):
- United States (24):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin